CLINICAL TRIAL: NCT06519695
Title: A Study on the Exercise Intervention Mode of Modern Exercises and Traditional Chinese Exercises for the Community-Dwelling Pre-frail Elderly: Based on the Wellness Motivation Theory
Brief Title: Exercise Intervention for Pre-frail Elderly
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Jianping Ren, director of department, Hangzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JRen
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Older Adults
Keywords: frail; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercises group (Experimental): Multicomponent exercise intervention under the guidance of the wellness motivation theory
  Interventions: Behavioral: Multicomponent exercises
- Control group (No Intervention): Health education about exercise only once.

INTERVENTIONS:
Behavioral: Multicomponent exercises — Performed exercise three times a week, one time at a community health service station and two times at home
  Arms: Multicomponent exercises group

SUMMARY:
The aim of this study is to evaluate the effectiveness of multicomponet exercise for reversing pre-frailty among Chinese community-dwelling pre-frail older adults.Meanwhile,to explore the effects of multicomponent exercise on self-efficiency of exercise.

DETAILED DESCRIPTION:
Based on the Wellness Motivation Theory (WMT), this study aimed to develop a theoretical model of exercise intervention for the pre-frail elderly. This study was to establish an exercise intervention mode, conduct empirical research through randomized controlled trials, and propose improvement strategies, aiming at improving the effectiveness of health management services for the community-dwelling pre-frail elderly. Specific research objectives are as follows:

1. To develop a theoretical model of exercise intervention for the pre-frail elderly based on the WMT, and to explain the operation mechanism of the exercise intervention mode.
2. An empirical study was conducted to verify the applicability and effectiveness of the exercise intervention mode, analyze the influencing factors of the intervention effect, and propose optimization strategies to improve the exercise intervention effect of the elderly in pre-frailty.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling prefrail older adults based on Fried frailty phenotype;
* age≥60 years,≤85 years;
* not engaged in regular physical activity or exercise programs in the previous 6 months;
* no hearing or visual impairment that might hinder communication;
* Written informed consent.

Exclusion Criteria:

* physical restrictions to perform the tests and/or exercises,
* cognitive impairment;
* medical contraindications for participation in an exercise program.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reversal of pre-frailty | 24 weeks
  Reversal rate of pre-frailty (from pre-frail to robust in this study)

SECONDARY OUTCOMES:
Self-efficacy for exercise | 24 weeks
  The Self-Efficacy for Exercise Scale was designed to test people's confidence to continue exercising despite barriers to exercise. The score of each item ranged from 0 to 10, with higher scores representing greater exercise self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Jianping, Principal Investigator — Hangzhou Normal University
Locations (1):
- Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dun Y, Hu P, Ripley-Gonzalez JW, Zhou N, Li H, Zhang W, Chen M, Zheng Q, Cui N, Wu S, Liu S. Effectiveness of a multicomponent exercise program to reverse pre-frailty in community-dwelling Chinese older adults: a randomised controlled trial. Age Ageing. 2022 Mar 1;51(3):afac026. doi: 10.1093/ageing/afac026. PMID 35231098
- [Result] McMahon SK, Wyman JF, Belyea MJ, Shearer N, Hekler EB, Fleury J. Combining Motivational and Physical Intervention Components to Promote Fall-Reducing Physical Activity Among Community-Dwelling Older Adults: A Feasibility Study. Am J Health Promot. 2016 Nov;30(8):638-644. doi: 10.4278/ajhp.130522-ARB-265. Epub 2016 Jun 16. PMID 26389979
- [Result] Barrachina-Igual J, Martinez-Arnau FM, Perez-Ros P, Flor-Rufino C, Sanz-Requena R, Pablos A. Effectiveness of the PROMUFRA program in pre-frail, community-dwelling older people: A randomized controlled trial. Geriatr Nurs. 2021 Mar-Apr;42(2):582-591. doi: 10.1016/j.gerinurse.2020.10.014. Epub 2020 Nov 12. PMID 33189414
- [Derived] Fang J, Ren J, Wang J, Qiu X, Zhang S, Yuan S, Wu L, Xie L. Combining motivational and exercise intervention components to reverse pre-frailty and promote self-efficacy among community-dwelling pre-frail older adults: a randomized controlled trial. BMC Geriatr. 2024 Oct 30;24(1):896. doi: 10.1186/s12877-024-05464-6. PMID 39478450